CLINICAL TRIAL: NCT04364256
Title: Neuromuscular Electrical Stimulation for Physical Function Maintenance During Hematopoietic Stem Cell Transplantation
Brief Title: Muscle Stimulation for Physical Function During Stem Cell Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: F3245-W; IK2RX003245-03 (NIH)
Record Dates: First submitted 2020-04-20; First posted 2020-04-28 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Autologous Hematopoietic Stem Cell Transplant
Keywords: neuromuscular electrical stimulation; physical function; hematologic cancer; muscle wasting; multiple myeloma; lymphoma; Hematopoietic Stem Cell Transplant; cancer cachexia; cancer rehabilitation
MeSH Terms: conditions — Hematologic Neoplasms; Muscular Atrophy; Multiple Myeloma; Lymphoma

STUDY DESIGN:
Intervention Model Description: Neuromuscular electrical stimulation (active vs sham signal)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: During Informed Consent, patients will be instructed to not presume group assignment. An unblinded study coordinator will then randomize each participant to NMES:Sham on a 1:1 basis, stratifying by diagnosis. The unblinded coordinator will ensure each participant performs the appropriate NMES or Sham stimulus on each training day; stimulation will only occur in private exam rooms. NMES and Sham stimulators will be outwardly identical apart from a concealed "A" or "B" label indicating NMES or Sham device; the designation of A or B will only be known to the unblinded study coordinator, and not to the PI. The PI will administer all outcome assessments and conduct all statistical analyses; therefore the PI will remain blinded to NMES vs Sham group assignment until study completion. In the study database, group assignment will be coded as A or B, the PI will not know the coding of A or B. A document containing the coding will be kept in a different electronic location than the study folder.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active NMES (Active Comparator): asymmetric biphasic waveforms at 71 pulses per second frequency (Hz), 400 s pulse duration, 5:10s on:off time (50% duty cycle), and 1.5s ramp-up time. Participants will be in control of the muscle stimulator devices at all times and will be instructed to perform all sessions in the supine position. Bilateral NMES will be delivered via asymmetric, biphasic using four cutaneous parallel channels delivered simultaneously using 2"x4" or 3"x5" self-adhesive electrodes. For the active NMES group, participants will be encouraged to increase the amplitude to a level of moderate discomfort, such as that experienced during conventional exercise, but not to induce pain. At minimum, the amplitude should induce visible muscle contraction.
  Interventions: Device: RS-4i Plus Sequential Stimulator (RS Medical, Vancouver, WA)
- Sham NMES (Sham Comparator): The amplitude of the muscle stimulators for the Sham group will be capped at 15 milliamperes so patients will only feel cutaneous sensation without achieving muscle contraction.
  Interventions: Device: RS-4i Plus Sequential Stimulator (RS Medical, Vancouver, WA)

INTERVENTIONS:
Device: RS-4i Plus Sequential Stimulator (RS Medical, Vancouver, WA) — Active or Sham Neuromuscular electrical stimulation. US Food and Drug Administration-approved 2012
  Other Names: NMES, e-stim

SUMMARY:
Some blood, bone marrow, and lymphatic (hematologic) cancers such as Hodgkin/Non-Hodgkin lymphomas, chronic lymphocytic leukemia, and multiple myeloma, are over-represented in Veterans due to exposures including Agent Orange and an increased percentage of patients of African American ethnicity. Hematologic transplantation (HCT) is a common treatment for these cancers, but often leads to deconditioning, fatigue, muscle atrophy, and poor quality of life, which are associated with complications such as hospitalization and infection. Despite the significance of these symptoms, there are no approved treatments to prevent/reverse these long-term effects. The cancer itself, side effects of chemotherapy, and sedentary behavior, contribute to these effects. Although exercise before and after HCT has helped reduce these effects, it is inconsistently recommended to patients and most remain sedentary through and after treatment. The investigators are testing an alternative exercise strategy, neuromuscular electrical stimulation, to maintain physical function quality of life after HCT.

DETAILED DESCRIPTION:
Hematopoietic cell transplantation (HCT) reduces physical function and muscle mass and increases fatigue. Neuromuscular electrical stimulation (NMES), when used as a stand-alone intervention, improves muscle strength and muscle mass in non-cancer patients with chronic obstructive pulmonary disease and chronic heart failure. The use of NMES to combat disuse atrophy and functional decline may be particularly useful in the HCT setting as patients undergo intensive preparatory chemotherapy and often experience symptoms including severe fatigue that leave them inactive or isolated for extended time periods surrounding the transplant. However, its use in the setting of cancer has not been well-established. This proposal will contribute to developing strategies toward optimizing the safety and outcomes associated with HCT in Veterans with hematologic malignancies. The overall goals of this study are to assess 1) the efficacy of an NMES vs Sham intervention on HCT-induced reductions in physical function and muscle mass and worsening of patient-reported fatigue and QOL and 2) the association between physical function and prolonged recovery of patient-reported fatigue and QOL. The investigators hypothesize that 1) NMES will attenuate the acute HCT-induced negative impact on physical function, body composition, QOL, and fatigue compared to Sham intervention, and 2) baseline physical function will be a significant predictor of 6-month recovery of patient-reported fatigue and QOL. Aim 1: To determine the efficacy of NMES vs. Sham for attenuation of HCT-induced reductions in physical function, muscle mass, and patient-reported QOL and fatigue in patients undergoing autologous HCT. Patients will be randomized 1:1 (NMES:Sham) stratified by diagnosis. Physical function, body composition, QOL, and fatigue will be assessed at baseline (Pre, after admission to the Bone Marrow Transplant Unit but before initiation of preparatory chemotherapy) and 28 plus or minus 5 days after HCT (Follow-up 1; FU1). The primary outcome will be between-group difference in 6MWT change at FU1 compared to Pre (N=23/group; 46 total). Secondary outcomes include: body composition measured by dual-energy x-ray absorptiometry; previously validated questionnaires (Functional Assessment of Chronic Illness Therapy-Fatigue; Muscle and Joint Measures) to assess patient-reported fatigue, QOL, symptom burden, and functional status; standard of care clinical/laboratory data regarding co-morbidities, adverse events, hospitalizations, treatment history, functional status, and clinical course; and NMES process measures such as feasibility, acceptability, adherence in number of sessions, accurate use, duration/intensity, complications, and satisfaction. Aim 2: To determine predictive ability of baseline 6MWT on delayed recovery of physical function, QOL, and fatigue, patient-reported outcomes, physical function, and chart review will be collected 6-months after HCT (FU2). 6MWT at Pre will be used to determine significant predictors of QOL and fatigue at FU2 (N=46) as assessed by previously validated questionnaires. Clinical measures extracted from medical charts will include changes from FU1 to FU2 in standard of care clinical/laboratory data regarding co-morbidities, adverse events, hospitalizations, functional status, treatment history, disease trajectory, and survival. Aim 3 (exploratory): To investigate the acute impact of NMES vs. Sham during HCT on various aspects of physical function and patient-reported QOL for determining potential endpoints for future clinical trials. Exploratory measures of function (stair climbing power; muscle strength; sit-to-stand; handgrip strength; peak oxygen consumption) assessed at Pre and FU1 will be used to determine significant predictors of exploratory QOL measures (Multidimensional Fatigue Inventory; Short Form-36; European Organization for Research and Treatment of Cancer QOL Questionnaire) assessed at FU2.

ELIGIBILITY:
Inclusion Criteria:

* adequate cognitive and language ability to provide consent
* Veteran enrolled in MTU at VAPSHCS for planned standard of care autologous HCT

Exclusion Criteria:

* active deep vein thrombosis or thrombophlebitis
* untreated hemorrhagic disorders
* concomitant study inclusion in other nutritional or physical exercise interventional trials
* concomitant use of anabolic agents
* rhabdomyolysis or other muscle conditions where NMES is contraindicated
* implanted cardiac device
* baseline patient-reported muscle soreness of 5-6 on the soreness likert scale that is unrelated to recent physical exertion
* history of prior hematologic stem cell transplant
* probable or definitive liver cirrhosis
* reduced renal clearance defined as Stage 4 chronic kidney disease (glomerular filtration rate <45 ml/min/1.73 m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-12-29 (Actual)

PRIMARY OUTCOMES:
6-Minute Walk Test | change from before to 1month after transplant
  Manual and mobile application assessment

SECONDARY OUTCOMES:
Patient-reported Fatigue | change from before to 1month after transplant
  Anderson Symptom Assessment Scale (range 0-10 where 10 is maximum fatigue)
Lean Body Mass | change from before to 1month after transplant
  dual energy fan-beam x-ray absorptiometry; bioelectrical impedance
Physical Activity | change from before to 1month after transplant
  triaxial accelerometry
NMES adherence | 1month after transplant
  Number of sessions completed out of total sessions
Muscle Damage (safety) | change from before to 2 weeks after intervention initiation
  plasma creatine kinase
Muscle Damage (safety) | change from before to 4 weeks after intervention initiation
  plasma creatine kinase
Muscle Damage (safety) | change from before to 6 weeks after intervention initiation
  plasma creatine kinase
Muscle Damage (safety) | change from before to 8 weeks after intervention initiation
  plasma creatine kinase
Muscle Damage (safety) | change from before to 1month after transplant
  plasma creatine kinase
6-Minute Walk Test | change from before to 6 months after transplant
  Mobile application assessment
Patient-reported Fatigue | change from before to 6 months after transplant
  Anderson Symptom Assessment Scale (range 0-10 where 10 is maximum fatigue)
Physical Activity | change from before to 6 months after transplant
  triaxial accelerometry

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey J Anderson, PhD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anderson LJ, Paulsen L, Miranda G, Syrjala KL, Graf SA, Chauncey TR, Garcia JM. Neuromuscular electrical stimulation for physical function maintenance during hematopoietic stem cell transplantation: Study protocol. PLoS One. 2024 May 10;19(5):e0302970. doi: 10.1371/journal.pone.0302970. eCollection 2024. PMID 38728244

DOCUMENTS (1):
  • Informed Consent Form (2023-09-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT04364256/ICF_000.pdf